CLINICAL TRIAL: NCT06712160
Title: Diagnostic Accuracy of Artificial Intelligence, CBCT, and Clinical Examination in Detecting Number of Root Canals in Conventional and Retreated Maxillary and Mandibular Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Misr International University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MIU-IRB-2425-008
Record Dates: First submitted 2024-11-21; First posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-10

CONDITIONS: Number of Root Canals
Keywords: CBCT; AI
MeSH Terms: interventions — Artificial Intelligence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CBCT, Clinical using DOM (Experimental): Comparing the three methods for the detection of the number of canals of maxillary and mandibular molars
  Interventions: Diagnostic Test: Artificial Intelligence

INTERVENTIONS:
Diagnostic Test: Artificial Intelligence — The number of canals detected by AI

SUMMARY:
The study compares the effectiveness of Artificial Intelligence (AI), CBCT, and clinical examination in detecting root canals in upper first, upper second, and lower first molars. Results show AI detects more molars with three or four canals in conventional treatment cases and retreatment cases.

DETAILED DESCRIPTION:
Introduction: Accurate root canal detection is crucial for successful endodontic treatment, particularly in complex molar cases. Conventional methods, such as clinical examination and cone-beam computed tomography (CBCT), have their limitations, as high radiation exposure. Recent advancements in Artificial Intelligence (AI) have shown promise in improving diagnostic accuracy. This study aims to compare the effectiveness of AI, CBCT, and clinical examination using a dental operating microscope (DOM) in detecting root canals in upper first, upper second, and lower first molars, in both conventional and retreatment cases. Methods: CBCT scans from 210 patients requiring non-surgical root canal therapy or re-treatment were selected. The scans were analyzed using three detection methods: clinical examination via DOM, interpretation by two experienced endodontists using CBCT, and an AI convolutional neural network (CNN) software (Diagnocat). The detected number of root canals was recorded and compared across the three methods.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients who were capable of providing informed consent
* Age between 18 to 40 years old.
* A restorable tooth.

Exclusion Criteria:

* Patients that underwent vital pulp therapies.
* Patients with calcifications in pulp space.
* Open apex/immature roots.
* Teeth restored by full coverage crowns.
* Pregnant women by taking adequate history from patient and pregnancy test that was done in the first visit

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 212 (Actual)
Dates: Start 2023-01-20 (Actual); Primary Completion 2024-01-20 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
The number of canals detected | 1 day
  The number of canals detected clinically using DOM, CBCT and by AI

SECONDARY OUTCOMES:
Canal Morphology | 1 day
  Canal morphology for successful and failed cases

CONTACTS AND LOCATIONS:
Locations (1):
- Misr International University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
will be shared after publishing the paper

DOCUMENTS (3):
  • Study Protocol (2024-10-29): https://cdn.clinicaltrials.gov/large-docs/60/NCT06712160/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-29): https://cdn.clinicaltrials.gov/large-docs/60/NCT06712160/SAP_001.pdf
  • Informed Consent Form (2024-10-29): https://cdn.clinicaltrials.gov/large-docs/60/NCT06712160/ICF_002.pdf